CLINICAL TRIAL: NCT01076985
Title: Special Investigation of Kaletra in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: PMOS-JAP-00-002
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2012-01-18 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2011-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lopinavir/ritonavir group: All pregnant women in this noninterventional, post-marketing observational study, who were prescribed lopinavir/ritonavir (Kaletra) in accordance with the local Prescribing Information for the treatment of HIV infection.
  Interventions: Drug: Lopinavir/ritonavir (Kaletra)

INTERVENTIONS:
Drug: Lopinavir/ritonavir (Kaletra) — Lopinavir/ritonavir (LPV/r) evaluated separately in patients who were naive to previous antiretroviral treatment and those who were not.
  Other Names: Lopinavir/ritonavir; Kaletra

SUMMARY:
This non-interventional, post-marketing observational study was conducted to obtain safety data from the use of lopinavir/ritonavir (Kaletra), in clinical practice, in pregnant women and their children in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who have received Kaletra for the treatment of HIV infection were eligible for this study

Exclusion Criteria:

* Contraindications according to the Package Insert:

  * Patients with a history of hypersensitivity to any ingredient of Kaletra
  * Patients who are receiving pimozide, cisapride, ergotamine tartrate, dihydroergotamine mesylate, ergometrine maleate, methylergometrine maleate, midazolam, triazolam, vardenafil hydrochloride hydrate, boriconazol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2000-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Maeda, Study Director — Abbott Japan Co.,Ltd
Locations (5):
- Japan (5):
  - Site Reference ID/Investigator# 35862, Aichi
  - Site Reference ID/Investigator# 35863, Okayama
  - Site Reference ID/Investigator# 35864, Osaka
  - Site Reference ID/Investigator# 35865, Tokyo
  - Site Reference ID/Investigator# 5326, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lopinavir/Ritonavir Group
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 24
Age Continuous [Median (Full Range); unit: years] | 30 [21 to 41]
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Region of Enrollment [Number; unit: participants]
  Japan | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Drug Reactions (ADRs)
Description: The number of patients (mothers and infants) with adverse drug reactions, defined as adverse events for which the causal relationship with Kaletra was something other than "not related" by the investigator (i.e., "probable," "possible," or "unclear"). ADRs are reported by preferred term and inclusive of all those reported at any visit. Although a patient may experience a particular preferred term more than once, each patient was counted only once for each preferred term.
Time Frame: During pregnancy and for one year after birth
Population: All available observed data for all participants and their resulting infants/live births are included.
Measure: Number; unit: participants
Groups:
- Lopinavir/Ritonavir: All pregnant women in this noninterventional, post-marketing observational study, who were prescribed lopinavir/ritonavir (Kaletra) in accordance with the local Prescribing Information for the treatment of HIV infection.
- Infants: Infants from live births of the pregnant women who were prescribed lopinavir/ritonavir (Kaletra) in accordance with the local Prescribing Information for the treatment of HIV infection and participated in this noninterventional, post-marketing observational study.
Arm/Group | Lopinavir/Ritonavir | Infants
Number analyzed (Participants) | 24 | 21
participants
  Anemia | 2 | 5
  Hypercholesterolemia | 1 | 0
  Hyperlipidemia | 1 | 0
  Diarrhea | 1 | 0
  Nausea | 2 | 0
  Rash | 1 | 1
  Abortion missed | 1 | 0
  Premature labor | 1 | 0
  Threatened labor | 1 | 0
  Neutropenia | 0 | 1
  Hypoglycemia | 0 | 1
  Cardio-respiratory arrest | 0 | 1
  Apnea | 0 | 1
  Neonatal respiratory distress syndrome | 0 | 1
  Transient tachypnea of the newborn | 0 | 1
  Small for dates baby | 0 | 1
  Pyrexia | 0 | 1

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during pregnancy and in their infants for up to one year after birth were reported.
Groups:
- Infants: Infants from live births of the pregnant women who were prescribed lopinavir/ritonavir (Kaletra) in accordance with the local Prescribing Information for the treatment of HIV infection who participated in this noninterventional, post-marketing observational study.
Arm/Group | Lopinavir/Ritonavir Group | Infants
Serious Adverse Events (participants affected / at risk) | 3/24 | 3/21
Other Adverse Events (participants affected / at risk) | 11/24 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir Group (N=24) | Infants (N=21)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature labor (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Threatened labor (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir Group (N=24) | Infants (N=21)
Anemia (Blood and lymphatic system disorders) | 6 | 10
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Breast enlargement (Reproductive system and breast disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Transient tachypnea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.